CLINICAL TRIAL: NCT00471978
Title: Molecular and Genetic Analysis of Lung Cancer
Brief Title: DNA Analysis of Blood and Tissue from Patients with Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Christopher Christiani, Elkan Blout Professor of Enviromental Genetics, Professor of Medicine, Massachusetts General Hospital
Other Study IDs: CDR0000450128; MGH-1999-P-004935/26 (Other: Partners Institutional Review Board)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; pulmonary carcinoid tumor
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help the study of cancer in the future.

PURPOSE: This clinical trial is analyzing the DNA in blood and tissue samples from patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the role of genetic polymorphisms in lung-cancer risk in patients with lung cancer.
* Assess the role of germline polymorphisms in DNA repair genes, p53 pathway genes, and a matrix metalloproteinase gene (tumor invasion factor) in lung-cancer risk, after adjusting for potential confounders.
* Assess the roles of gender and age in the genetic susceptibility of lung cancer.
* Assess the role of genetic polymorphisms in modifying the diet-lung cancer risk association (gene-diet and exploratory gene-gender-diet and gene-gene-diet interactions).
* Assess the role of polymorphisms on the risk of developing specific histologic subtypes of lung cancer in case-only analyses.
* Determine whether continued exposures to mainstream and/or second-hand tobacco smoking is associated with poorer clinical prognosis in patients treated for lung cancer.

OUTLINE: This began as a case-control study, but is currently case only.

Blood samples are collected from patients and controls. Samples are analyzed by polymerase chain reaction for gene polymorphisms. Genes to be studied include GSTP1, GSTM1, GSTT1, ERCC2, XRCC1, EPHX, NAT-2, p53 gene, CYP1A1, NQO1, MnSOD, and GPX1. Tissue samples collected from patients undergoing surgery and blood samples are archived for future studies.

Patients and controls complete questionnaires about diet, medical history, and occupational/environmental history.

PROJECTED ACCRUAL: A total of 3,400 patients and 3,400 controls will be accrued for early phases of this study. Total enrollment to reach 15,000.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient:

  * Newly diagnosed primary lung cancer

    * Patient at Massachusetts General Hospital (MGH) or Boston Medical Center Cancer Center

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

EXCLUSIONS:

Vulnerable populations are excluded. Patients with metastasis from another site to lung or mesothelioma are excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Metabolic polymorphisms | 10 years
  to compare differences among lung cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: David C. Christiani, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard School of Public Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No